CLINICAL TRIAL: NCT00400829
Title: A Phase 2 Study of the Halichondrin B Analog E7389 in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC) Previously Treated With a Taxane
Brief Title: E7389 in Treating Patients With Recurrent or Progressive Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01159; NCI-2009-01159 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000514516; PHII-74 (Other: City of Hope); 7437 (Other: CTEP); N01CM62204 (NIH); N01CM62201 (NIH); N01CM62209 (NIH)
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Results first posted 2015-01-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2013-10

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — eribulin

ARMS (1):
- Arm I (Experimental): Patients receive 1.4 mg/m2 eribulin mesylate IV over 1-2 minutes on days 1 and 8. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: eribulin mesylate

INTERVENTIONS:
Drug: eribulin mesylate — Given IV
  Other Names: B1939; E7389; ER-086526; halichrondrin B analog

SUMMARY:
This phase II trial is studying how well E7389 works in treating patients with recurrent or progressive stage IIIB or stage IV non-small cell lung cancer. Drugs used in chemotherapy, such as E7389, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Evaluate the antitumor activity of E7389 (eribulin mesylate), in terms of objective response rate, in patients with recurrent or progressive stage IIIB or IV non-small cell lung cancer.

II. Evaluate the time to progression and overall survival of patients treated with this drug.

III. Evaluate the toxicity profile of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive eribulin mesylate IV over 1-2 minutes on days 1 and 8. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed once monthly for at least 6 months and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)
* Stage IIIB or IV disease
* Recurrent or progressive disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* Must have received prior treatment with platinum-based therapy and a taxane
* Asymptomatic brain metastasis allowed provided off steroids for > 2 weeks
* Zubrod performance status (PS) ≤ 2 OR Karnofsky PS 60-100%
* Life expectancy > 3 months
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 2.0 mg/dL
* AST/ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No neuropathy ≥ grade 2
* No uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would preclude study compliance
* No other concurrent investigational agents
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* At least 2 weeks since prior radiotherapy, including palliative radiotherapy, and recovered
* No more than 2 prior chemotherapy regimens for NSCLC in the metastatic or adjuvant setting
* No concurrent combination antiretroviral therapy for HIV-positive patients

Exclusion Criteria:

* Absolute neutrophil count ≥ 1,500/mm³
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to E7389

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gitlitz, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I
Started | 66
Completed | 66
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 66
Age, Continuous [Median (Full Range); unit: years] | 63 [35 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 66

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (CR or PR) According to RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT, MRI or X-ray: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Tumor measurements repeated every 6 weeks
Measure: Number; unit: percentage of patients responding
Arm/Group | Arm I
Number analyzed (Participants) | 66
percentage of patients responding | 5

2. Secondary Outcome: Overall Survival
Description: Will be estimated using the product-limit method of Kaplan and Meier.
Time Frame: From start of treatment to death from any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I
Number analyzed (Participants) | 66
Months | 11.6 [8.2 to 13.7]

3. Secondary Outcome: Progression Free Survival
Description: Will be estimated using the product-limit method of Kaplan and Meier.
Time Frame: From start of treatment to the time of documented progression, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I
Number analyzed (Participants) | 66
Months | 2.7 [1.3 to 3.9]

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded over a 40 month period.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Groups:
- Arm I: Patients receive eribulin mesylate IV over 1-2 minutes on days 1 and 8. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  eribulin mesylate: Given IV
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 23/66
Other Adverse Events (participants affected / at risk) | 65/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=66)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 2 (2)
Disease progression (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Leukocyte count decreased (Investigations) | 2 (3)
Leukopenia (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 13 (19)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=66)
Hemoglobin decreased (Blood and lymphatic system disorders) | 46 (159)
Cardiac disorder (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (4)
Hearing loss (Ear and labyrinth disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 1 (1)
Extraocular muscle paresis (Eye disorders) | 1 (3)
Eye disorder (Eye disorders) | 1 (2)
Vision blurred (Eye disorders) | 3 (4)
Watering eyes (Eye disorders) | 2 (7)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 10 (14)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 17 (29)
Diarrhea (Gastrointestinal disorders) | 7 (18)
Dyspepsia (Gastrointestinal disorders) | 7 (11)
Dysphagia (Gastrointestinal disorders) | 2 (3)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 8 (10)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 16 (28)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (8)
Chest pain (General disorders) | 9 (14)
Chills (General disorders) | 2 (4)
Death (General disorders) | 11 (11)
Disease progression (General disorders) | 30 (30)
Edema limbs (General disorders) | 11 (25)
Fatigue (General disorders) | 45 (137)
Fever (General disorders) | 9 (14)
Gait abnormal (General disorders) | 1 (1)
General symptom (General disorders) | 4 (14)
Injection site reaction (General disorders) | 1 (2)
Localized edema (General disorders) | 1 (6)
Pain (General disorders) | 7 (10)
Hepatic pain (Hepatobiliary disorders) | 2 (4)
Bronchitis (Infections and infestations) | 5 (5)
Catheter related infection (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (14)
Paranasal sinus infection (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 2 (3)
Sinusitis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Activated partial thromboplastin time prolonged (Investigations) | 1 (2)
Alanine aminotransferase increased (Investigations) | 11 (31)
Alkaline phosphatase increased (Investigations) | 12 (43)
Aspartate aminotransferase increased (Investigations) | 15 (25)
Bilirubin increased (Investigations) | 5 (5)
Creatinine increased (Investigations) | 2 (3)
Forced expiratory volume decreased (Investigations) | 1 (1)
INR increased (Investigations) | 2 (7)
Laboratory test abnormal (Investigations) | 2 (4)
Leukocyte count decreased (Investigations) | 38 (147)
Leukopenia (Investigations) | 4 (6)
Lymphocyte count decreased (Investigations) | 27 (104)
Neutrophil count decreased (Investigations) | 38 (126)
Platelet count decreased (Investigations) | 7 (10)
Serum cholesterol increased (Investigations) | 2 (4)
Weight loss (Investigations) | 4 (6)
Anorexia (Metabolism and nutrition disorders) | 24 (49)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 4 (7)
Blood glucose increased (Metabolism and nutrition disorders) | 31 (84)
Dehydration (Metabolism and nutrition disorders) | 4 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 20 (48)
Serum calcium decreased (Metabolism and nutrition disorders) | 6 (7)
Serum calcium increased (Metabolism and nutrition disorders) | 6 (8)
Serum glucose decreased (Metabolism and nutrition disorders) | 4 (5)
Serum magnesium decreased (Metabolism and nutrition disorders) | 5 (10)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 7 (13)
Serum potassium decreased (Metabolism and nutrition disorders) | 9 (13)
Serum potassium increased (Metabolism and nutrition disorders) | 4 (6)
Serum sodium decreased (Metabolism and nutrition disorders) | 12 (23)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (37)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (10)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 7 (20)
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 8 (22)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (8)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (26)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (22)
Acoustic nerve disorder NOS (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (7)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 11 (15)
Headache (Nervous system disorders) | 10 (15)
Neuralgia (Nervous system disorders) | 1 (2)
Neurological disorder NOS (Nervous system disorders) | 2 (3)
Peripheral motor neuropathy (Nervous system disorders) | 2 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 27 (67)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Taste alteration (Nervous system disorders) | 2 (7)
Tremor (Nervous system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 6 (20)
Confusion (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 5 (8)
Insomnia (Psychiatric disorders) | 6 (9)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (3)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 3 (4)
Urethral pain (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (13)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 5 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (56)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 22 (70)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (54)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (7)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 6 (7)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2)
Flushing (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 3 (6)
Phlebitis (Vascular disorders) | 1 (5)
Thrombosis (Vascular disorders) | 1 (6)
Vascular disorder (Vascular disorders) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less